CLINICAL TRIAL: NCT06026592
Title: Detection of Plasma DNA of Renal Origin in Kidney Transplant Patients
Acronym: DART-REIN
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230298
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury; Renal Transplantation
Keywords: Epigenetic; Renal cell-free DNA; Transplantation; biomarkers
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: determination of circulating biomarkers of renal origin circulating biomarkers of renal origin — The extracted circulating DNA will be extracted and converted using the methylation kit. Finally, circulating DNA will be analyzed using the PCR mix developed by CGenetix, quantifying tubular and glomerular biomarkers (patented technology).

SUMMARY:
Donor-derived cell-free DNA (dd-cfDNA) has been proposed as a potential diagnostic tool to monitor the rejection status of the kidney transplant. It has been suggested that dd-cfDNA is increasing in the blood of kidney transplant patient presenting a graft rejection. In this project, investigators proposed a different approach to predict and characterize kidney transplant rejection/dysfunction based on the quantification of epigenetic signatures present on the donor-cell-free DNA. In 2018, Moss et al. develops a deconvolution model capable of identifying the tissue origin of circulating DNA by taking advantage of its epigenetic properties. The study confirmed that the cell-free DNA circulating in healthy subjects comes mainly from blood cells and endothelial cells, but not from kidney cells.

In this study, researchers investigate the evolution of blood renal-specific cell-free DNA amount in patient with chronic kidney disease before and after the transplantation surgery by testing a set of renal-specific epigenetic markers. The purpose of this study is to identify the biological noise of "native kidney" on renal-specific cell-free DNA and to compare it with signal coming from "transplanted kidney".

DETAILED DESCRIPTION:
At the diagnostic level, routine monitoring of graft functionality after kidney transplantation relies on the use of non-specific markers, such as serum creatinine (allowing estimation of glomerular filtration rate or GFR) and proteinuria. Definitive diagnosis of renal allograft dysfunction still requires invasive allograft biopsy, which remains the gold standard for assessing graft status. The histopathological diagnosis of renal graft dysfunction is based on the Banff classification and makes it possible to examine the immune infiltrate and the cellular lesions of the graft to make a precise diagnosis. However, Renal biopsy has certain limitations: 1/ It is invasive for the patient, with associated complications, mainly hemorrhagic in 1 to 3.5% of cases; 2/ Its effectiveness in predicting early rejection (3 months) post-transplant remains controversial. A lack of patient benefit has been proven by several studies for screening biopsy; 3/ Histological analysis is subject to intra- and inter-observer variations; and 4/ it is an expensive examination due to the medical time required to perform and interpret the biopsy.

The "donor-cell-free DNA (dd-cfDNA)" has been suggested as a diagnostic tool at the service of the graft. Analyzes based on molecular signatures on the circulating DNA of the donor (Single Polymorphism Nucleotide (SNP)) have made it possible to discriminate the circulating cell-free DNA from the transplanted kidney (from the donor) from the circulating cell-free DNA specific to the recipient. Data from several studies suggest that blood dd-cfDNA levels can detect rejection in heart, lung, liver and kidney allografts. First studied by multiplex qPCR and then NGS technologies, the SNPs present on the dd-cfDNA were then quantified by digital PCR techniques.

In this study, investigators proposed a different approach to predict and characterize kidney transplant rejection/dysfunction based on the quantification of epigenetic signatures present on the donor-cell-free DNA. In 2018, Moss et al. develops a deconvolution model capable of identifying the tissue origin of circulating DNA by taking advantage of its epigenetic properties. The study confirmed that the cell-free DNA circulating in healthy subjects comes mainly from blood cells and endothelial cells, but not from kidney cells. In 2023, Loyfer et al. proposed a methylation atlas of more than 200 cells type and suggested that each cell has its own epigenetic signature that can be study in cell-free DNA.

In this study, researchers investigate the evolution of blood renal-specific cell-free DNA amount in patient with chronic kidney disease before and after the transplantation surgery by testing a set of renal-specific epigenetic markers. The purpose of this study is to identify the biological noise of "native kidney" on renal-specific cell-free DNA and to compare it with signal coming from "transplanted kidney". Researchers hypothesize that the biological noise from "native kidney" in chronic kidney diseases is negligible compared to that of the post-transplantation graft.

To investigate this hypothesis, investigators collect blood samples before and after transplant surgery to quantify kidney-specific cell-free DNA markers. They also proposed to quantify cell-free DNA markers of graft perfusion fluid to validate the specificity of renal markers and to study graft tissue damage during organ transport. Each renal-cell-free DNA sample is quantified by a proprietary technologies using a multiplex digital-PCR assay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* With end-stage renal failure
* Summoned for a kidney transplant at Pitié Salpêtrière Hospital
* Having been informed of the study and not objecting to the study having given free and informed written consent for the genetic analysis
* Benefiting from a social security scheme (excluding AME)

Exclusion Criteria:

Under legal protective measures (curatorship or guardianship, under judicial safeguard).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with end-stage renal disease about to receive a kidney transplant from a deceased donor.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
Amount of renal circulating cell-free DNA | 6 hours before kidney transplantation and 12 to 24 after transplantation surgery
  The amount of renal-cell-free DNA (glomerular and tubular markers) will be measured 6 hours before the kidney transplant is performed and 12-24 hours after the kidney transplant by digital multiplex PCR

SECONDARY OUTCOMES:
Estimating the inter-individual variations of the free circulating methylome of renal origin in patients with end-stage chronic insufficiency | 6 hours before kidney transplantation and 12 to 24 after transplantation surgery
  The amount of renal-cell-free DNA (glomerular and tubular markers) measured will be compared between individuals.
Identify by a method without a priori (methyl seq) specific markers of acute renal injury in terms of epigenetic signature | 6 hours before kidney transplantation and 12 to 24 after transplantation surgery
  Comparison of two biomarkers quantification methods (whole genome methyl-Sequencing and multiplex digital-PCR)
Study the statistical association between the presence of free circulating methylated sequences of renal origin and the resumption of graft function | 7 day after the transplant
  Comparison of circulating free methylome of renal origin between the groups of patients with immediate recovery of function and delayed recovery of function (defined on the performance of a dialysis session in the first 7 days and on the reduction ratio serum creatinine between the 1st and 2nd day after the transplant).

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié-Salpétriêre Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.